CLINICAL TRIAL: NCT05371223
Title: Combined Nabpaclitaxel Pressurized IntraPeritoneal Aerosol Chemotherapy With Systemic Nabpaclitaxel-Gemcitabine Chemotherapy for Pancreatic Cancer Peritoneal Metastases - A Single-arm, Open-label, Phase II Trial: Nab-PIPAC Trial
Brief Title: Combined Nabpaclitaxel Pressurized IntraPeritoneal Aerosol Chemotherapy With Systemic Nabpaclitaxel-Gemcitabine Chemotherapy for Pancreatic Cancer Peritoneal Metastases
Acronym: Nab-PIPAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4368
Record Dates: First submitted 2022-03-16; First posted 2022-05-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Peritoneal Carcinomatosis; Pancreas Neoplasm
MeSH Terms: conditions — Peritoneal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Experimental): Eligible patients affected by pancreatic cancer PM will be enrolled according to in-/exclusion criteria.
  Each patient will be scheduled for three treatment combined courses for a total of six cycles of endovenous Nabpaclitaxel-Gemcitabine chemotherapy and three of Nabpaclitaxel-PIPAC.
  Interventions: Drug: Combined Nabpaclitaxel Pressurized IntraPeritoneal Aerosol Chemotherapy With Systemic Nabpaclitaxel-Gemcitabine

INTERVENTIONS:
Drug: Combined Nabpaclitaxel Pressurized IntraPeritoneal Aerosol Chemotherapy With Systemic Nabpaclitaxel-Gemcitabine — Each combined course is constituted by two consecutive 28-day cycles of systemic chemotherapy (three adminstrations per cycle: days 1,8 and 15) and one cycle of PIPAC administered within 10-13 days from the last administration of systemic chemotherapy. Between each combined course a 7-10 days pause is observed.
  The recommended dose of Nabpaclitaxel in combination with Gemcitabine is 125 mg/m2 administered endovenous over 30 minutes on Days 1, 8 and 15 of each 28-day cycle. The concurrent recommended dose of Gemcitabine is 1000 mg/m2 administered intravenously over 30 minutes immediately after the completion of Nabpaclitaxel administration on Days 1, 8 and 15 of each 28-day cycle.
  A pressurized aerosol containing Nabpaclitaxel at the dose of 112,5 mg/m2 diluted in a total volume of 200 ml of NaCl 0.9% is applied through the nebulizer inside the abdominal cavity during laparoscopy.

SUMMARY:
Combined chemotherapy consisting of endovenous Nabpaclitaxel-Gemcitabine and Nabpaclitaxel-PIPAC may be a promising treatment for patients affected by pancreatic cancer PM who are in need of curative options.

The purpose of this study is to evaluate the antitumoral activity of combined Nabpaclitaxel-PIPAC and systemic Nabpaclitaxel-Gemcitabine chemotherapy for pancreatic cancer peritoneal metastases.

Secondary objectives include the evaluation of the feasibility, the safety, further assessment of the antitumoral activity, the overall and progression free survival, the QoL, the pharmacokinetics of Nabpaclitaxel PIPAC.

Furthermore, the study aims to evaluate the patients' nutritional status and the molecular evolution of PM along treatment with a time-course translational research.

DETAILED DESCRIPTION:
Pancreatic carcinoma (PC) is an aggressive neoplasm carrying a high metastatic potential with a 5-year survival rate of 7%. The vast majority of cases already developed locally advanced disease, and distant metastases are present at the time of diagnosis. Furthermore, the recurrence rate is nearly 80% within the first two years after surgery, and about half of these patients show peritoneal relapse. Palliative systemic chemotherapy represents the standard treatment option in case of peritoneal metastases (PM) from PC but roughly reaches a median overall survival of 6-11 months with more than 5% of serious adverse events.

Based on the available data, Nabpaclitaxel is indicated in combination with Gemcitabine for the first-line systemic treatment of patients with metastatic adenocarcinoma of the pancreas.

Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) is a novel intraperitoneal drug-delivery system of low-dose chemotherapy as a pressurized aerosol. Until now, the combination cisplatin/doxorubicin or oxaliplatin has been administered by PIPAC. Recently, a phase I study (NCT03304210) was conducted to explore the use of intraperitoneal Nabpaclitaxel administered by PIPAC, confirming its safety and preliminary efficacy. The recommended dose to safely start a phase-II study was 112.5 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Willing and able to provide written and informed consent;
* Histological or cytological proof of pancreatic cancer;
* Metastatic disease with peritoneal carcinomatosis determined by the treating physician, based on abdominal CT or MR and/or diagnostic laparotomy or laparoscopy;
* Evaluable disease defined by RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* Life expectancy of at least 3 months;
* No contraindication for laparoscopy;
* No contraindication for drugs used in the study;
* Adequate bone marrow function: Absolute neutrophil count ≥ 1500 cell./mm3; Platelets ≥ 100000 cell./mm3;
* Hemoglobin ≥ 9 g/dl
* Adequate renal function (serum creatinine up to 1.5 times the maximal limit of the local laboratory) or else based upon clinical evaluation;

Exclusion Criteria:

* Advanced metastatic systemic disease with clinical deterioration;
* Patients with extraabdominal tumor spread;
* Patients with a germline or somatic pathogenic variant involving an (Homologous Recombination Repair) HRR-related gene;
* Symptoms of gastrointestinal occlusion and total parenteral nutritional support;
* Patients defined as "refractory" to previous systemic treatment with Nab-paclitaxel and Gemcitabine administered for locally advanced pancreatic cancer (patients treated with Nabpaclitaxel-Gemcitabine for a locally advanced disease may be included if PM developed after at least 6 months from the end of previous chemotherapy);
* History of severe and unexpected reactions to Nabpaclitaxel or Gemcitabine derivates
* Known hypersensitivity reaction to drugs chemically related to Nabpaclitaxel, Gemcitabine and their excipients;
* Severe cardiac disease (recent myocardial ischemia, severe cardiac arrhythmias, severe cardiac failure);
* Clinical disease progression after first 2 months of systemic Nabpaclitaxel Gemcitabine chemotherapy;
* Any concurrent severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk of associated with study participation or investigational product administration or may interfere with compliance with study procedures or the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | Three and a half years
  The Disease Control Rate (DCR) defined as the combined incidence of complete response (CR), partial response (PR) and stable disease (SD) according to the RECIST v. 1.1 criteria during study treatments and the EOT visit.

SECONDARY OUTCOMES:
The compliance to treatment | Three and a half years
  - The number of patients unable to undergo six cycles of systemic chemotherapy combined with three PIPAC cycles and reasons for discontinuation.
Toxicity assessed by CTCAE | Three and a half years
  * The number of patients with major toxicity, defined as grade ≥3 according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0 during the on-study evaluation phase and up to 4 weeks after the last chemotherapy administration.
  * The number of patients with minor toxicity, defined as grade ≤2 according to CTCAE v5.0 during the treatment period and up to 4 weeks after the last chemotherapy administration.
Postoperative complication assessed by Clavien-Dindo | Three and a half years
  -The number of patients with major and minor postoperative complications, defined as grade ≥3 and grade ≤2 according to Clavien-Dindo, respectively, during the treatment period and up to 4 weeks after the last PIPAC procedure.
Antitumoral activity assessed by PRGS | Three and a half years
  -The pathological tumor response, based on the review of peritoneal biopsies collected during each PIPAC, performed by a pathologist blinded to clinical outcomes using the Peritoneal Regression Grading Score (PRGS). A patient will be considered a responder if any reduction in the PRGS during subsequent biopsies will be recorded;
  (PRGS 1: Complete regression without cancer cells - PRGS 2: higher response with prevalence of regressive phenomena and only a few residual cancer cells - PRGS 3: minor response with prevalence of residual cancer cells and poor regressive phenomena - PRGS 4: no response to therapy without regressive phenomena A reduction in the PRGS during subsequent biopsies will be considered as a positive response.)
Antitumoral activity assessed by PCI | Three and a half years
  -The macroscopic tumor response, based on Peritoneal Cancer Index (PCI) recorded during each PIPAC;
  The PCI index will be calculated according to the Sugarbaker method, which provides the assignment of a score between 0 and 3 based on the size of peritoneal metastases (0 without lesions; 1 if diam. 0.5 cm; 2 if diam. between 0.5 and 5 cm; 3 if diam > 5 cm or coalescent lesions) observed in 12 regions of the peritoneal cavity. The maximum score is 39.
Antitumoral activity assessed by ascites volume | Three and a half years
  - The macroscopic tumor response, based on ascites volume recorded during each PIPAC
Antitumoral activity assessed by tumor markers | Three and a half years
  - The biochemical tumor response, based on tumor markers (CEA, Ca 19.9, Ca 125) measured at different time points.
The Progression Free Survival (PFS) | From treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  the time between treatment start and one of the following events, whichever comes first:
  * radiologic progression based on RECIST criteria v. 1.1,
  * clinical progression (eg, bowel occlusion, inability to oral feeding, refractory ascites),
  * death;
The Overall Survival (OS) | From treatment start to death, assessed up to 12 months
  The Overall Survival (OS) is defined as the time between treatment start and death.

OTHER OUTCOMES:
The intravenous area under the curve (AUC) of paclitaxel | Three and a half years
  The concentration of paclitaxel in peritoneal samples. The penetration of paclitaxel in peritoneal tissues.
Intra-patient e intra-tumoral heterogeneity | Three and a half years
  - The germline mutational profile from blood samples
Identification of pancreatic cancer disease evolution trough pathway analysis a in primary tumor and peritoneal sites during treatments | Three and a half years
  - The genomic mutational profile of PM biopsies taken during PIPAC;

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Di Giorgio, MD, Principal Investigator — UOS trattamenti integrati della carcinosi peritoneale avanzata -UOC Chirurgia del peritoneo e retroperitoneo - Fondazione Policlinico Universitario A. Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Giorgio A, Ferracci F, Bagala C, Carbone C, Salvatore L, Strippoli A, Attalla El Halabieh M, Abatini C, Alfieri S, Pacelli F, Tortora G. Combined Nabpaclitaxel pressurized intraPeritoneal aerosol chemotherapy with systemic Nabpaclitaxel-Gemcitabine chemotherapy for pancreatic cancer peritoneal metastases: protocol of single-arm, open-label, phase II trial (Nab-PIPAC trial). Pleura Peritoneum. 2024 Nov 6;9(3):121-129. doi: 10.1515/pp-2024-0010. eCollection 2024 Sep. PMID 39544430